CLINICAL TRIAL: NCT04799444
Title: Complications Post COVID-19 - Observational Study in Children and Adults
Brief Title: LATE-COVID/LATE-COVID-Kids - Observational Study in Children and Adults
Acronym: LATE-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Maciej Banach, MD,PhD,FNLA,FAHA,FESC,FASA, Polish Mother Memorial Hospital Research Institute
Other Study IDs: LATE-COVID
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID-19; post-COVID-19; late-COVID-19 complications; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The study is planned also to be extended with the genetic predisposition in children to COVID-19 late complications (within independent grant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients with complications post COVID-19
- Children with complications post COVID-19

SUMMARY:
All consecutive patients admitted to the Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland between 1st October 2020 and 31st December 2021 due to symptoms, which might reflect complications following COVID-19, will be included in the observational cohort study. Data concerning clinical characteristics, results of laboratory tests, other studies, such as: echocardiography, 24 hours ambulatory ECG recording will be collected. The study is planned also to be extended with the genetic predisposition in children to COVID-19 late complications (within independent grant).

DETAILED DESCRIPTION:
A wide range of complications have been linked to COVID-19 - the coronavirus disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). It is well known that COVID-19 affects multiple organs. Most of the data however present the early complications during the acute phase of the infection, and there is still a lack of knowledge on the late complications that might appear after recovery. Additionally, the long-term complications in patients who were asymptomatic or had mild symptoms during the acute phase of infection, not requiring hospitalization, oxygen therapy or mechanical ventilation has not been fully studied. Therefore, our aim was to assess factors related to the severity of post-COVID complications among patients without severe symptoms in the acute phase of COVID-19. The study will include consecutive COVID-19 convalescents (the infection of coronavirus was confirmed with real-time polymerase chain reaction test or positive result of autoantibodies) admitted to the Departments of Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland, for complications. Both children and adults will be included in the study. The patients will have laboratory testing and other studies due to the character of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* consecutive COVID-19 convalescents (the infection of coronavirus was confirmed with real-time polymerase chain reaction test or positive result of autoantibodies) admitted to the Departments of Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland, for complications

Exclusion Criteria:

* no history of COVID-19 infection,
* lack of complications post COVID-19,
* severe course of Sars-COV-2 infection,
* lack pf patient's agreement to be included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive COVID-19 convalescents admitted to the Departments of Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland, for complications
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe post-COVID-19 complications | Baseline
  Data concerning clinical characteristics, results of laboratory tests, other studies, such as: echocardiography, 24 hours ambulatory ECG recording will be collected. According to the results patients will be qualified to severe or mild complication group
Factors related to the severity of post-COVID-19 complications | Baseline
  Data concerning clinical characteristics, results of laboratory tests, other studies, such as: echocardiography, 24 hours ambulatory ECG recording will be collected to verify which of them can be related to the severity of post-COVID-19 complications.

OTHER OUTCOMES:
Post-COVID SCORE | Baseline
  We aim to create a post-COVID SCORE that helps to predict the risk of late complications both in children and adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Polish Mother Memorial Research Institute (PMMHRI) in Lodz, Poland, Lodz, Poland

REFERENCES:
- [Background] Parsamanesh N, Karami-Zarandi M, Banach M, Penson PE, Sahebkar A. Effects of statins on myocarditis: A review of underlying molecular mechanisms. Prog Cardiovasc Dis. 2021 Jul-Aug;67:53-64. doi: 10.1016/j.pcad.2021.02.008. Epub 2021 Feb 20. PMID 33621589
- [Background] Petrovic V, Radenkovic D, Radenkovic G, Djordjevic V, Banach M. Pathophysiology of Cardiovascular Complications in COVID-19. Front Physiol. 2020 Oct 9;11:575600. doi: 10.3389/fphys.2020.575600. eCollection 2020. PMID 33162899
- [Background] Bhaskar S, Sinha A, Banach M, Mittoo S, Weissert R, Kass JS, Rajagopal S, Pai AR, Kutty S. Cytokine Storm in COVID-19-Immunopathological Mechanisms, Clinical Considerations, and Therapeutic Approaches: The REPROGRAM Consortium Position Paper. Front Immunol. 2020 Jul 10;11:1648. doi: 10.3389/fimmu.2020.01648. eCollection 2020. PMID 32754159
- [Background] Radenkovic D, Chawla S, Pirro M, Sahebkar A, Banach M. Cholesterol in Relation to COVID-19: Should We Care about It? J Clin Med. 2020 Jun 18;9(6):1909. doi: 10.3390/jcm9061909. PMID 32570882
- [Result] Lewek J, Jatczak-Pawlik I, Maciejewski M, Jankowski P, Banach M. COVID-19 and cardiovascular complications - preliminary results of the LATE-COVID study. Arch Med Sci. 2021 Mar 18;17(3):818-822. doi: 10.5114/aoms/134211. eCollection 2021. PMID 34025853